CLINICAL TRIAL: NCT04045808
Title: Associate Professor
Brief Title: Relationship of Oral Status to Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Collaborators: Ankara University (Other)
Responsible Party: Principal Investigator, Mehtap Bilgin Çetin, PhD,DDS, Baskent University
Other Study IDs: Cetin
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Coronary Artery Disease; Periodontal Diseases
Keywords: coronary angiography; coronary artery disease; edentulism; periodontitis; periodontal disease
MeSH Terms: conditions — Coronary Artery Disease; Periodontal Diseases; Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CAD(+) group: Participants were included in CAD (+) if they had more than 50% reduction in diameter in one or more major epicardial arteries,
  Interventions: Other: radiographic evaluations were done
- CAD(-) group: patients with less than 50% reduction in epicardial artery diameter were enrolled to CAD (-) group
  Interventions: Other: radiographic evaluations were done

INTERVENTIONS:
Other: radiographic evaluations were done — For radiographic analysis, periapical radiographs were taken from teeth with ≥ 4mm PPD using a hand held intra-oral x-ray system operating at 60kVp, 1.5 mA . The alveolar bone loss was measured by a personal computer with the Microsoft Windows XP operating system with original software.

SUMMARY:
We hypothesized that periodontal disease and edentulism could be a risk for CAD and there might be a relationship between the oral status and the number of main coronary vessels with ≥ 50% stenosis. Therefore, primary goal of this study is to investigate the connection between oral status and the extent of coronary artery disease (CAD), which is diagnosed by angiography.

DETAILED DESCRIPTION:
Subjects were grouped as CAD (+) or CAD (-) based on their coronary angiography outcomes. Participants were included in CAD (+) if they had more than 50% reduction in diameter in one or more major epicardial arteries, whereas patients with less than 50% reduction in epicardial artery diameter were enrolled to CAD (-) group.The extent of CAD was measured by the number of main coronary vessels with more than 50% stenosis and occluded left main coronary artery (LMCA) was also noted.Demographic and socioeconomic backgrounds, brushing and interdental cleaning habits, frequency of dental visits, levels of education and medical histories of participants were carefully recorded. Medical histories mainly included cardiovascular risk factors consisting of age, gender, family history of heart disease and myocardial infarction (MI), smoking habits, current medications, body mass index (BMI), hypertension, diabetes, high density protein (HDL) and CRP levels. BMIs of participants were obtained through dividing weight (in kilograms) by the square of height (in meters). Blood samples were collected before angiography in order to analyze biological parameters. Hospital records were consulted to obtain patient information such as existence of hypertension, hyperlipidemia, and diabetes mellitus. Education levels were evaluated based on the last school the patient had graduated from and categorized as no education, secondary school, high school and university.During the examination, remaining teeth count, plaque index (PI), gingival index (GI), bleeding on probing (BOP) and probing pocket depth (PPD) were analyzed. Periodontal measurements were recorded at four sites around each tooth (mesial, mid-buccal, distal, and mid-lingual) by a periodontal probe excluding third molars. Each patient was evaluated for PI, GI, PPD average scores (whole-mouth) and percent of BOP (+) sites. Oral status was categorized in three groups: Group 1 consisted of periodontally healthy subjects and patients with gingivitis. Patients having periodontitis were involved in group 2 and group 3 included edentulous subjects. Periodontal health was defined as the absence of gingivitis or periodontitis. Gingivitis was defined as BOP score of ≥ 10% and probing depth of ≤ 3mm. Diagnosis of periodontitis is based on multiple clinical and radiographic parameters. If a patient has one or more sites of inflammation (BOP), ≥ 2mm radiographic bone loss and ≥ 4mm probing depth; he/she will be diagnosed for periodontitis.

For radiographic analysis, periapical radiographs were taken from teeth with ≥ 4mm PPD using a hand held intra-oral x-ray system operating at 60kVp, 1.5 mA by Dexcowin DX 3000 with a CCD based sensor Trophy RVG ver. 5.0 . The alveolar bone loss was measured by a personal computer with the Microsoft Windows XP operating system with original software. The site where periodontal ligament terminates at the surface of the root was labeled as the alveolar bone crest. Apart from the third molars, all teeth were examined to measure the interval between cementoenamel junction and interproximal alveolar crest, regarding both mesial and distal aspects of each tooth.

ELIGIBILITY:
Inclusion Criteria:patients who were admitted to Ankara University, Faculty of Medicine, Department of Cardiology and had coronary angiography.

Exclusion Criteria:Participants who needed antibiotic prophylaxis before the dental examination, had periodontal treatment or used antibiotics during the last 6 months were excluded from the study, along with the pregnant women.

Ages: 30 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: who were admitted to Ankara University, Faculty of Medicine, Department of Cardiology and had coronary angiography
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2009-04-12 (Actual); Primary Completion 2011-01-01 (Actual); Study Completion 2011-02-02 (Actual)

PRIMARY OUTCOMES:
Oral status of patients | Oral status of a patient was defined in 20 minutes.
  Oral status was categorized in three groups: Group 1 consisted of periodontally healthy subjects and patients with gingivitis. Patients having periodontitis were involved in group 2 and group 3 included edentulous subjects. Periodontal health was defined as the absence of gingivitis or periodontitis. Gingivitis was defined as BOP score of ≥ 10% and probing depth of ≤ 3mm. Diagnosis of periodontitis is based on multiple clinical and radiographic parameters. If a patient has one or more sites of inflammation (BOP), ≥ 2mm radiographic bone loss and ≥ 4mm probing depth; he/she will be diagnosed for periodontitis

SECONDARY OUTCOMES:
medical histories of participants | Medical data was recorded in 20 minutes
  Medical histories mainly included cardiovascular risk factors consisting of age, gender, family history of heart disease and myocardial infarction (MI), smoking habits, current medications, body mass index (BMI), hypertension, diabetes.BMIs of participants were obtained through dividing weight (in kilograms) by the square of height (in meters).Hospital records were consulted to obtain patient information such as existence of hypertension, hyperlipidemia, and diabetes mellitus. If the patient was taking medication for hyperlipidemia, he was noted as a patient with hyperlipidemia.If the patient was taking medication for diabetes, he was noted as a patient with diabetes.If the patient was taking medication for hypertension, he was noted as a patient with hypertension.according to smoking status, patients divided into three groups as never smoked, current smokers, former smokers.